CLINICAL TRIAL: NCT01476072
Title: 31P MRS Ischaemic Exercise Optimisation and COPD Myopathy Study
Brief Title: 31P MRS Ischaemic Exercise Optimisation and COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 113784
Record Dates: First submitted 2011-09-29; First posted 2011-11-22 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Atrophy, Muscular
MeSH Terms: conditions — Muscular Atrophy | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no treatment (No Intervention): MRI scans only
  Interventions: Other: MRI scan

INTERVENTIONS:
Other: MRI scan — MRI scan only, methodology study with no other intervention

SUMMARY:
An MRI study to develop a reliable methodology for 31P MRS ischaemic exercise in order to obtain a consistent standard of measurement of muscle metabolism while maintaining an acceptable level of subject comfort and use optimised method to measure and compare metabolism in the biceps and quadriceps of patients with COPD-related myopathy and control subjects

DETAILED DESCRIPTION:
31P Magnetic Resonance Spectroscopy (31P MRS) is a non-invasive method to measure muscle metabolism during exercise. This protocol is intended to provide information for planning future clinical trials applying 31P MRS as an endpoint measure for proof of pharmacology studies with novel therapeutic molecules. Parts A & B of this study will refine imaging and exercise protocols for 31P MRS during brief periods of muscle ischaemia and will assess the test-retest variance. In Part C we will apply 31P MRS with aerobic exercise in a pilot study to estimate differences in skeletal muscle oxidative metabolism between age- and sex-matched control subjects and patients with myopathy associated with Chronic Obstructive Pulmonary Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Fit to safely tolerate procedures
2. Male or female between 18 and 80 years of age
3. If pre-menopausal female, non-pregnant on dipstick urinalysis
4. Subject and responsible physician agree that the subject will be able to comfortably lie in scanning position in the scanner for up to 90 minutes
5. Capable of giving written informed consent
6. All four limbs are intact and free of disease

The following criteria apply to patients with COPD myopathy only:

1. Established diagnosis of COPD with a disease classification of GOLD Stage II and above with suspected or established diagnosis of myopathy and/or COPD with low BMI (under 20 for men and under 19 for women) and/or MVC under 120% of the BMI.
2. At least a 20 pack year history of smoking
3. Resting oxygen saturation above 85% on room air
4. Ambulant and not oxygen-dependent at rest or during mild exertion

Exclusion Criteria:

1. Ineligible for MRI/MRS scanning in accordance to local MR safety regulations
2. Any medical condition, acute or chronic, that will lead to potential discomfort when lying supine in the magnet for periods up to 90 min
3. Any medical condition that will lead to potential discomfort with repetitive movement of the limb being tested in the scanner
4. Subjects undergoing ischaemic/anaerobic 31P MRS must have no history of clinically significant peripheral vascular disease, abnormal blood clotting, deep vein thrombosis or pulmonary embolism or suspected clinically significant signs of limb vascular disease on screening examination.
5. Subjects undergoing ischaemic/anaerobic 31P MRS must not have taken the oral contraceptive pill, hormone replacement therapy, or undergone anaesthesia within past 1 month, or have a history of recent prolonged immobility greater than 4 hours (e.g. air travel), or considered unfit in the opinion of the study physician
6. Concurrent medical conditions known or suspected that in the opinion of the responsible physician could confound interpretation of results.
7. A medical or psychiatric history that in the opinion of the responsible physician would risk safety of the subject or well-being of the subject.

The following criteria apply to control subjects and COPD patients participating in Part C of the study:

1. Oxygen saturations below 85% on room air at rest, or significant desaturation on mild exertion.
2. Current or recent (<4 weeks) infectious exacerbation of COPD requiring corticosteroid therapy at the time of screening or scanning visit day.
3. Any significant medical illness other than COPD which, in the opinion of the study physician, may preclude participation or which by virtue of being associated with muscle weakness may cause distortion of the results (e.g. neuromuscular disease, severe heart failure &c).
4. Control subjects with any history of regular smoking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
level of skeletal muscle metabolism | 1 year
  ADP, ATP, PCr, Pi, and pH will be measured during rest, anaerobic exercise and recovery to determine muscle metabolism.

SECONDARY OUTCOMES:
determine Markers of disease in patients with COPD-related myopathy | 1 year
  tests such as spirometry, muscle biopsy, muscle cross-sectional area CSA, muscle strength to indicate level of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, London, United Kingdom